CLINICAL TRIAL: NCT02943915
Title: The WISE Trial - Walking Improvement for SCI With Exoskeleton
Acronym: WISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ekso Bionics (Industry)
Collaborators: Burke Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105333
Record Dates: First submitted 2016-09-27; First posted 2016-10-25 (Estimated); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Injuries, Spinal Cord
Keywords: Spinal Cord; Injury; Exoskeleton; Ekso; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Wounds and Injuries | interventions — Exoskeleton Device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Group 1: Ekso GT Rehabilitation Therapy (Experimental): Participants in this group receive Ekso GT (gait training) PT therapy intervention 3 times per week for 12 weeks (36 sessions). Intervention: Ekso GT Rehabilitation therapy
  Interventions: Device: Ekso GT Rehabilitation Therapy
- Group 2: Active controls - BWSTT Therapy (Active Comparator): Participants in this group receive a matched number of sessions of standard gait training using body-weight supported treadmill training and overground training. Intervention: Body Weight Supported Treadmill Training
  Interventions: Device: Body Weight Supported (BWS) Treadmill Training
- Group 3: Passive controls (No Intervention): Participants in this group continue with normal daily activities over 12 weeks.

INTERVENTIONS:
Device: Ekso GT Rehabilitation Therapy — Walking Improvement for Spinal Cord Injuries with Exoskeleton
  Other Names: Exoskeleton
  Arms: Group 1: Ekso GT Rehabilitation Therapy
Device: Body Weight Supported (BWS) Treadmill Training — Standard gait training using BWS PT and overground training
  Other Names: Conventional Therapy
  Arms: Group 2: Active controls - BWSTT Therapy

SUMMARY:
A randomized, controlled trial comparing exoskeleton gait training with standard gait training or no gait training in community-dwelling participants with chronic incomplete spinal cord injury

DETAILED DESCRIPTION:
Community dwelling iSCI participants may improve clinical gait function by engaging in a gait training regimen, where robotic exoskeletons can readily deliver a precise dose and simultaneously reduce the physical stress imposed on therapists using conventional manually assisted stepping practice. Exoskeleton training is predicted to improve function in participants receiving usual care, but not superior to intensity-matched manual training. The rationale to implement exoskeleton robotics as preference in gait training is based on precision dosing, over-ground training, and reduced therapist burden for high repetition training.

The investigators aim to demonstrate that Ekso exoskeleton training can significantly improve gait speed in stable chronic, community-dwelling incomplete SCI (iSCI) participants. The objectives of this study are the following:

A. Primary Objective:

To demonstrate that a 12 week robotic gait training regimen can lead to a clinically meaningful improvement in independent gait speed on the 10 Meter Walk Test (10MWT) in community dwelling participants with chronic iSCI.

B. Secondary Objectives:

1. To examine the economic factors such as number of physical therapists/staff required during training.
2. To analyze the physical burden on therapists assisting and supervising during training.
3. To study the influence of factors that may modify the gait recovery in the chronic incomplete SCI population (demographic, clinical, functional, psychological, balance, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Motor incomplete paraplegia or tetraplegia
2. Neurological level of injury (NLI) C1- approximately T10 (inclusive, for upper motor neuron injuries only), as determined by the International Standards for Neurological Classification of SCI (ISNCSCI)
3. Sufficient diaphragmatic strength such that respiration is not compromised with exercise.
4. Sufficient upper extremity strength to use a front wheeled walker either by manual muscle testing (minimum triceps strength bilaterally of 3/5, shoulder abduction/adduction and flexion/extension 4/5)
5. AIS-C SCI & AIS-D SCI, as determined by the International Standards for Neurological Classification of SCI (ISNCSCI)
6. Ambulates at <0.44 meters/second with or without physical assistance and assistance device
7. WISCI ≥ 1
8. 18 - 75 yrs, inclusive
9. No current or history of other neurological conditions
10. Screened and cleared by a physician
11. Involved in standing program or must be able to tolerate at least 15 min upright
12. Weigh 220 pounds (100kg) or less
13. Be able to fit into the Ekso device
14. Approximately between 5'0" and 6'4" tall
15. Standing hip width of approximately 18" or less
16. Have near normal range of motion in hips, knees and ankles

Exclusion Criteria:

1. AIS-A SCI or AIS-B SCI
2. Lower motor neuron injuries, as shown by absent reflexes during bilateral quadriceps and Achilles tendon taps
3. < 3 months since previous intensive gait training regimen
4. Already walking at self-selected ambulation speeds of at least 0.44 meter/second with or without assistance
5. Currently involved in another intervention study
6. Concurrent neurological disease
7. Hip flexion contracture greater than ~17°
8. Knee flexion contracture greater than 12°
9. Unable to achieve neutral ankle dorsiflexion with passive stretch (neutral with max 12° knee flexion)
10. Leg length discrepancy

    1. Greater than 0.5" for upper leg
    2. Greater than 0.75" for lower leg
11. Spinal instability
12. Unresolved deep vein thrombosis
13. Uncontrolled autonomic dysreflexia
14. Severe muscular or skeletal pain
15. Spasticity that prevents joint motion (severe stiffness or rigidity,) where both legs have a Modified Ashworth Score (MAS) score of 3 or higher for half or more of their proximal lower extremity muscles; proximal muscles include hip flexors/extensors/adductors and knee flexors/extensors.
16. Open skin ulcerations on buttocks or other body surfaces in contact with exoskeleton or harness
17. Pregnancy
18. Cognitive impairments - unable to follow 2 steps commands and communicate for pain or to stop session
19. Shoulder extension Range of Motion (ROM) < 50° excludes crutches during sit to stand or vice versa. (Walking with crutches permitted.)
20. Participant requires the assistance of more than one therapist to transfer safely.
21. Uncontrolled or severe orthostatic hypotension that limits standing tolerance; defined as sustained, symptomatic drops in systolic and diastolic blood pressure when moving from sitting to standing
22. Active heterotrophic ossification (HO), hip dysplasia or hip/knee axis abnormalities
23. Colostomy
24. History of long bone fractures since the SCI, secondary to osteoporosis
25. Unable to sustain current medication regimen
26. Any reason the physician may deem as harmful to the participant to enroll or continue in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-09; Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Edwards, PhD, Principal Investigator — Burke Medical Research Institute
Locations (10):
- United States (10):
  - Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Gaylord Hospital, Wallingford, Connecticut
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Marianjoy Rehabilitation Hospital, Wheaton, Illinois
  - Kennedy Kruger Institute, Baltimore, Maryland
  - Rehabilitation Institute of Michigan, Detroit, Michigan
  - Courage Kenny Research Center, Minneapolis, Minnesota
  - Kessler Foundation, West Orange, New Jersey
  - Burke Medical Research Institute, White Plains, New York
  - TIRR Memorial Hermann Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stampacchia G, Rustici A, Bigazzi S, Gerini A, Tombini T, Mazzoleni S. Walking with a powered robotic exoskeleton: Subjective experience, spasticity and pain in spinal cord injured persons. NeuroRehabilitation. 2016 Jun 27;39(2):277-83. doi: 10.3233/NRE-161358. PMID 27372363
- [Background] Gad PN, Gerasimenko YP, Zdunowski S, Sayenko D, Haakana P, Turner A, Lu D, Roy RR, Edgerton VR. Iron 'ElectriRx' man: Overground stepping in an exoskeleton combined with noninvasive spinal cord stimulation after paralysis. Annu Int Conf IEEE Eng Med Biol Soc. 2015 Aug;2015:1124-7. doi: 10.1109/EMBC.2015.7318563. PMID 26736463
- [Background] Kozlowski AJ, Bryce TN, Dijkers MP. Time and Effort Required by Persons with Spinal Cord Injury to Learn to Use a Powered Exoskeleton for Assisted Walking. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):110-21. doi: 10.1310/sci2102-110. Epub 2015 Apr 12. PMID 26364280
- [Background] Kressler J, Thomas CK, Field-Fote EC, Sanchez J, Widerstrom-Noga E, Cilien DC, Gant K, Ginnety K, Gonzalez H, Martinez A, Anderson KD, Nash MS. Understanding therapeutic benefits of overground bionic ambulation: exploratory case series in persons with chronic, complete spinal cord injury. Arch Phys Med Rehabil. 2014 Oct;95(10):1878-1887.e4. doi: 10.1016/j.apmr.2014.04.026. Epub 2014 May 17. PMID 24845221
- [Background] Sale P, Russo EF, Russo M, Masiero S, Piccione F, Calabro RS, Filoni S. Effects on mobility training and de-adaptations in subjects with Spinal Cord Injury due to a Wearable Robot: a preliminary report. BMC Neurol. 2016 Jan 28;16:12. doi: 10.1186/s12883-016-0536-0. PMID 26818847
- [Background] Kolakowsky-Hayner SA, Crew J, Moran S, Shah A. Safety and feasibility of using the EksoTM bionic exoskeleton to aid ambulation after spinal cord injury. Spine. 2013 doi.org/10.4172/2165-7939.S4-003
- [Background] Forrest GF, Hutchinson K, Lorenz DJ, Buehner JJ, Vanhiel LR, Sisto SA, Basso DM. Are the 10 meter and 6 minute walk tests redundant in patients with spinal cord injury? PLoS One. 2014 May 1;9(5):e94108. doi: 10.1371/journal.pone.0094108. eCollection 2014. PMID 24788068

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Run-in category arm contains participants that began the intervention protocol to ensure that assessment and training procedures were practiced and followed as required in the clinical trial protocol. Following the satisfactory completion of at least one set of midpoint assessments during the run-in phase, subsequent main study participants (a separate cohort) were enrolled and randomly assigned. Run-in participant data was not collected or included in these results.
Groups:
- Run-in: Panients in this group began the intervention protocol for the EksoGT group to ensure that assessment and training procedures were practiced and followed as required in the clinical trial protocol.
Period: Overall Study
Arm/Group | Group 1: Ekso GT Rehabilitation Therapy | Group 2: Active Controls - BWSTT Therapy | Group 3: Passive Controls | Run-in
Started | 14 | 13 | 6 | 12
Completed | 9 | 10 | 6 | 12
Not Completed | 5 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0 | 0
Not completed — excluded | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants in the EksoGT run-in trial were for the learning of the therapists carrying out study protocol. While these participants were trained on the EksoGT, further data was not collected and no data was analyzed, including baseline characteristics. These numbers also do not include participants who withdrew from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ekso GT Rehabilitation Therapy | Group 2: Active Controls - BWSTT Therapy | Group 3: Passive Controls | Total
Number analyzed (Participants) | 12 | 12 | 6 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 5 | 27
  >=65 years | 0 | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 41.67 [26 to 58] | 51.91 [28 to 71] | 49 [26 to 74] | 47.2 [26 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 1 | 12
  Male | 7 | 6 | 5 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 6 | 30
Time since injury [Mean (Standard Deviation); unit: years] | 8.40 (8.59) | 7.04 (4.37) | 4.37 (4.77) | 7.05 (6.49)

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Speed From Baseline to 12 Weeks Using 10 Meter Walk Test (10MWT)
Description: The mean change in gait speed demonstrated during the 10MWT after 12 weeks of training and compared between groups. Positive values indicate improvement in gait speed (faster) from baseline to 12 weeks. Negative values indicate a reduction in gait speed (slower) from baseline to 12 weeks.
Time Frame: Baseline and 12 Weeks
Population: Population does not include participants who withdrew, who did not have completed outcome data, who were excluded, or who were included in the Ekso protocol run-in. Run in participants did not have data collected on them and were only utilized to to ensure that assessment and training procedures were practiced and followed as required in the clinical trial protocol.
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Group 1: Ekso GT Rehabilitation Therapy | Group 2: Active Controls - BWSTT Therapy | Group 3: Passive Controls
Number analyzed (Participants) | 9 | 10 | 6
meters/second | 0.18 (0.23) | 0.07 (0.11) | 0.03 (0.03)

2. Secondary Outcome: Number of Participants Who Met the Minimal Clinically Important Difference of 0.15m/s in Gait Speed Per 10 Meter Walk Test (10MWT) From Baseline to 24 Weeks
Description: Number of participants who achieve the Minimal Clinically Important Difference (MCID) of 0.15 m/s during the 10MWT when comparing between baseline gait speed and gait speed at 24 weeks.
Time Frame: Between baseline and 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ekso GT Rehabilitation Therapy | Group 2: Active Controls - BWSTT Therapy | Group 3: Passive Controls
Number analyzed (Participants) | 9 | 10 | 6
Participants | 3 | 2 | 0

3. Secondary Outcome: Change in Distance Covered Over 6 Minutes From Baseline to 24 Weeks
Description: 6 minute walk test (6MWT) completed at baseline and 24 weeks. Change assessed. Positive values indicate an increase in distance was able to be walked at 24 weeks versus at baseline. Negative values indicate a decrease in distance was walked at 24 weeks versus at baseline.
Time Frame: Baseline-24 weeks
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: feet
Arm/Group | Group 1: Ekso GT Rehabilitation Therapy | Group 2: Active Controls - BWSTT Therapy | Group 3: Passive Controls
Number analyzed (Participants) | 9 | 10 | 6
feet | 538 [268 to 687.3] | 346.6 [219.5 to 711.5] | 320 [148.8 to 466.6]

4. Secondary Outcome: Change in Time Required to Complete Timed Up and Go (TUG) Test From Baseline to 24 Week Follow up
Description: Examined balance and walking in participants at baseline and follow up at 24 weeks. Positive values indicate an improvement of time (less time) required to complete task at 24 week follow up versus at baseline. Negative values indicate a decline, more time required to complete task at follow up versus baseline.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: seconds
Arm/Group | Group 1: Ekso GT Rehabilitation Therapy | Group 2: Active Controls - BWSTT Therapy | Group 3: Passive Controls
Number analyzed (Participants) | 9 | 10 | 6
seconds | 26.4 [17.3 to 53] | 30 [26 to 70.7] | 46 [29 to 64.9]

5. Secondary Outcome: Number of Participants Who Experienced a Fall During Protocol
Description: At each training session, assessed if participant had experienced any falls. Count is number of participants who reported that yes, they did experience a fall.
Time Frame: Throughout 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ekso GT Rehabilitation Therapy | Group 2: Active Controls - BWSTT Therapy | Group 3: Passive Controls
Number analyzed (Participants) | 9 | 10 | 6
Participants | 0 | 0 | 0

6. Secondary Outcome: Change in Berg Balance Scale Score From Baseline to 24 Weeks
Description: Measurement of static and dynamic sitting and standing balance completed at baseline and at 24 weeks. Berg balance scale is a 14 item test with each item scored from 0-4. Possible scores range from 0-56. Higher scores indicate a lower risk of falls and better balance. Positive numbers indicate an improvement in Berg balance scale (scored out of 56), meaning that the participant scored higher at 24 weeks than at baseline. Negative values indicate a decline in performance of the Berg balance scale (scored out of 56), meaning that the participant scored lower at 24 weeks than at baseline.
Time Frame: Baseline-24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: Ekso GT Rehabilitation Therapy | Group 2: Active Controls - BWSTT Therapy | Group 3: Passive Controls
Number analyzed (Participants) | 12 | 11 | 6
score on a scale | 18.7 (10.4) | 19.22 (8.4) | 17.3 (6.5)

ADVERSE EVENTS:
Time Frame: AEs tracked through each participant's intervention period over 12 consecutive weeks.
Description: Participants using devices, no risk for death
Groups:
- Ekso Run in Participants: Participants in this group receive Ekso GT (gait training) PT therapy intervention but were not included in full data collection. This was completed to help the therapists get used to the protocol and use of the device.
Arm/Group | Group 1: Ekso GT Rehabilitation Therapy | Group 2: Active Controls - BWSTT Therapy | Group 3: Passive Controls | Ekso Run in Participants
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/13 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 12/14 | 9/13 | 3/6 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ekso GT Rehabilitation Therapy (N=14) | Group 2: Active Controls - BWSTT Therapy (N=13) | Group 3: Passive Controls (N=6) | Ekso Run in Participants (N=12)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | NA
lower extremity numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
allergic reaction to medication (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ekso GT Rehabilitation Therapy (N=14) | Group 2: Active Controls - BWSTT Therapy (N=13) | Group 3: Passive Controls (N=6) | Ekso Run in Participants (N=12)
Blood pressure issues (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Increased blood pressure resulting in treatment cessation
Fall (Musculoskeletal and connective tissue disorders) | 4 (12) | 5 (14) | 1 (4) | 4 (9) — Participant experienced any type of fall (from standing, from seated position) in or outside of any therapy treatment
Illness (Infections and infestations) | 5 (6) | 2 (4) | 0 (0) | 3 (3) — Illnesses including flu, common cold, stomach virus, nausea, bronchitis, prostate infection
Nerve pain or numbness (Nervous system disorders) | 2 (4) | 1 (1) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 6 (8) | 0 (0) | 4 (9) — included musculoskeletal pain, headache, and internal organ pain
Planned medical or surgical procedure (Surgical and medical procedures) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Skin bruising, redness, or rash (Skin and subcutaneous tissue disorders) | 6 (9) | 3 (4) | 0 (0) | 3 (5)
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (4) | 4 (7) | 2 (2) | 0 (0) — UTI

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT02943915/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT02943915/SAP_001.pdf
  • Informed Consent Form (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT02943915/ICF_002.pdf